CLINICAL TRIAL: NCT07176533
Title: Opioid-Free Pediatric Tonsillectomy With Intraoperative Maxillary Nerve Block Via Suprazygomatic Injection (OPTIMaS): A Randomized Controlled Triple-Blinded Trial
Brief Title: Suprazygomatic Maxillary Nerve Block in Pediatric Tonsillectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Abhijit Biswas, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SZMN inTonsillectomy
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Tonsillitis
Keywords: Pain control; Tonsillectomy; Adenotonsillectomy; Suprazygomatic maxillary nerve block; Anesthesia
MeSH Terms: conditions — Tonsillitis; Agnosia

STUDY DESIGN:
Intervention Model Description: Single-center prospective randomized controlled trial of suprazygomatic maxillary nerve block with placebo for pediatric patient undergoing tonsillectomy or adenotonsillectomy.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprazygomatic maxillary nerve block (SZMN) with bupivacaine (Experimental): Participants will receive 15 mg/kg of Tylenol and 6 mg/kg of celecoxib (a nonsteroidal anti-inflammatory (NSAID drug) up to a maximum dose of 200 mg prior to the start of general anesthesia which will consist of gas or intravenous induction (2 mcg/kg fentanyl, 0.5 mg/kg dexamethasone). The SZMN block will be performed using 0.2 ml/kg bilaterally of 0.25% bupivacaine (MARCAINE) (cumulative dose 0.4 ml/kg) (local anesthetic), up to a maximum dose of 5 mL per side. The surgery (tonsillectomy or adenotonsillectomy) will then proceed according to standard of care practices.
  Interventions: Procedure: Suprazygomatic maxillary nerve block (SZMN) with bupivacaine
- Suprazygomatic maxillary nerve block (SZMN) with placebo (Placebo Comparator): Participants will receive 15 mg/kg of Tylenol and 6 mg/kg of celecoxib (a nonsteroidal anti-inflammatory (NSAID drug) up to a maximum dose of 200 mg prior to the start of general anesthesia. which will consist of gas or intravenous induction (2 mcg/kg fentanyl, 0.5 mg/kg dexamethasone). The SZMN block will be performed using 0.2 ml/kg of saline (placebo) up to a maximum dose of 5 mL per side. The surgery (tonsillectomy or adenotonsillectomy) will then proceed according to standard of care practices.
  Interventions: Procedure: Suprazygomatic maxillary nerve block (SZMN) with placebo

INTERVENTIONS:
Procedure: Suprazygomatic maxillary nerve block (SZMN) with bupivacaine — Participants will receive 15 mg/kg of Tylenol and 6 mg/kg of celecoxib (a nonsteroidal anti-inflammatory (NSAID drug) up to a maximum dose of 200 mg prior to the start of general anesthesia which will consist of gas or intravenous induction (2 mcg/kg fentanyl, 0.5 mg/kg dexamethasone). The SZMN block will be performed using 0.2 ml/kg bilaterally of 0.25% bupivacaine (MARCAINE) (cumulative dose 0.4 ml/kg) (local anesthetic), up to a maximum dose of 5 mL per side. . The surgery (tonsillectomy or adenotonsillectomy) will then proceed according to standard of care practices.
  Arms: Suprazygomatic maxillary nerve block (SZMN) with bupivacaine
Procedure: Suprazygomatic maxillary nerve block (SZMN) with placebo — Participants will receive 15 mg/kg of Tylenol and 6 mg/kg of celecoxib (a nonsteroidal anti-inflammatory (NSAID drug) up to a maximum dose of 200 mg prior to the start of general anesthesia. which will consist of gas or intravenous induction (2 mcg/kg fentanyl, 0.5 mg/kg dexamethasone). The SZMN block will be performed using 0.2 ml/kg of saline (placebo) up to a maximum dose of 5 mL per side. The surgery (tonsillectomy or adenotonsillectomy) will then proceed according to standard of care practices.
  Arms: Suprazygomatic maxillary nerve block (SZMN) with placebo

SUMMARY:
Tonsillectomies are among the most common surgical procedures performed in pediatric populations, with more than 14,000 procedures performed annually in Ontario, with more than 80% being performed to treat sleep-disordered breathing, including sleep apnea. Despite being a routine procedure, postoperative pain is a prevalent challenge following tonsillectomies, with significant pain lasting 7 to 10 days and peaking within the first 3 days following surgery. Effective pain management is critical not only to enhance patient comfort, but to ensure functional recovery, decrease the risk of post-surgical complications, and reduce the risk of hospital readmissions. The suprazygomatic maxillary nerve block (SZMN block) has become a promising alternative to opioids for the management of post-tonsillectomy pain. The SZMN block numbs the nerves in the facial region that would contribute to feeling pain following tonsillectomy. Although the SZMN block has been successful in adult tonsillectomies and pediatric cleft palate repairs, its success in pediatric tonsillectomies remains under investigation. This randomized controlled trial aims to evaluate the efficacy and safety of the SZMN block in pediatric tonsillectomy and adenotonsillectomy patients, through its role in providing pain management over 14 days following surgery. This study will be conducted at Victoria Hospital, London Health Sciences Centre.

DETAILED DESCRIPTION:
Tonsillectomies are among the most common surgical procedures performed in pediatric populations, with more than 14,000 procedures performed annually in Ontario. Despite being a routine procedure, postoperative pain is a prevalent challenge following tonsillectomies, with significant pain lasting 7 to 10 days and peaking within the first 3 days following surgery. Effective pain management is critical not only to enhance patient comfort, but to ensure functional recovery, decrease the risk of post-surgical complications, and reduce the risk of hospital readmissions. More than 80% of tonsillectomies are performed to treat sleep-disordered breathing (SDB), an array of conditions including obstructive sleep apnea (OSA) that are characterized by abnormal respiratory patterns during sleep. Patients with these conditions often undergo an upregulation of central μ-opioid receptors due to chronic apnea, decreasing their response to hypercarbia and increasing opioid sensitivity. When opioids are administered for pain management, these patients are at a greater risk of hypoventilation and hypoxemia. Many nonopioid analgesics such as acetaminophen, non-steroidal anti-inflammatory drugs, and some corticosteroids provide varying degrees of efficacy in pain relief, acting more effectively in combination with other medications to maximize pain management while mitigating adverse effects.

The suprazygomatic maxillary nerve block (SZMN block) has become a promising alternative to systemic opioids for the management of post-tonsillectomy pain. The SZMN block targets the palatine branch of the maxillary nerve in the pterygopalatine fossa, providing partial analgesia to the adenoids while avoiding the glossopharyngeal nerve, thereby preserving airway reflexes and reducing the risk of respiratory compromise. Although the SZMN block has been successful in adult tonsillectomies and pediatric cleft palate repairs, its success in pediatric tonsillectomies remains under investigation. Reported complications are rare and easily managed, including perioperative bleeding and postoperative hematoma formation at the injection site. A recent randomized clinical trial by Lin et al. demonstrated the efficacy of the SZMN block in reducing opioid use and alleviating postoperative pain in pediatric patients during the immediate postoperative period, particularly the post-anesthesia care unit (PACU) stay and the first three days following surgery. However, its efficacy in pediatric tonsillectomy patients has not been evaluated over the initial 14-day postoperative period, during which patients commonly experience sustained, significant pain. The current investigation aims to evaluate the efficacy and safety of the SZMN block in pediatric tonsillectomy and adenotonsillectomy patients, through its role in providing pain management over 14 days following surgery.

Prior to enrollment in the study, informed consent will be sought from the parents/guardians of these children and assent will be obtained where appropriate. Upon enrollment in the study, patients will be randomized by a computer generated sequence into one of two study groups. The investigators, participants, and outcome assessors will be blinded to participant group assignment at the time of randomization and throughout treatment and assessment.

Group 1: Participants will receive 15 mg/kg of Tylenol and 6 mg/kg of celecoxib (a nonsteroidal anti-inflammatory (NSAID drug) up to a maximum dose of 200 mg prior to the start of general anesthesia which will consist of gas or intravenous induction (2 mcg/kg fentanyl, 0.5 mg/kg dexamethasone). The SZMN block will be performed using 0.2 ml/kg bilaterally of 0.25% bupivacaine (MARCAINE) (cumulative dose 0.4 ml/kg) (local anesthetic), up to a maximum dose of 5 mL per side. The surgery (tonsillectomy or adenotonsillectomy) will then proceed according to standard of care practices.

Group 2: Participants will receive 15 mg/kg of Tylenol and 6 mg/kg of celecoxib (a nonsteroidal anti-inflammatory (NSAID drug) up to a maximum dose of 200 mg prior to the start of general anesthesia. which will consist of gas or intravenous induction (2 mcg/kg fentanyl, 0.5 mg/kg dexamethasone). The SZMN block will be performed using 0.2 ml/kg of saline (placebo) up to a maximum dose of 5 mL per side. The surgery (tonsillectomy or adenotonsillectomy) will then proceed according to standard of care practices.

SZMN Block: Participants will lie in the supine position, and anatomical landmarks including the posterior orbital rim and the zygomatic arch will be identified and marked. The skin will be prepared with chlorhexidine gluconate 2% in isopropyl alcohol 70%. The Pajunk SonoBlock II needle will be inserted between the angle made by the posterior orbital rim and zygomatic arch until contacting the greater wing of the sphenoid bone. The needle alignment will be adjusted obliquely forward and caudally to access the pterygopalatine fossa, and negative aspiration will be confirmed. Study group participants will receive 0.2 ml/kg of 0.25% bupivacaine, to a maximum dose of 5 ml per side, deposited on the maxillary bone surface. Control group participants will receive 0.2 ml/kg of saline, to a maximum dose of 5 ml, deposited on the maxillary bone surface.

Following the completion of surgery, participants will be transferred to the post-anesthesia care unit (PACU) for recovery. While in the PACU, participants will be assessed at two different time points for opioid consumption, side effects, recovery progress, and for early postoperative pain. Pain will be assessed using the FLACC (Face, Legs, Activity, Cry, Consolability) Pain Scale.. This scale is a validated pain assessment tool that allows for assessment of pain in children. Scores for each category are assigned on a scale of 0-2 and then added together to receive a final pain score out of 10 which is then interpreted to determine the severity of pain the patient is experiencing where 0 indicates no pain and 10 indicates severe pain.

After the participant is discharged from the hospital, the study team will call the participants' parents/guardians on days 1, 7, and 14 following surgery to conduct a phone follow up visit. During each phone call, parents/guardians will be asked to answer questions about their child's pain, side effects, ability to swallow, opioid use, other medications that are being taken, pain rating, and parental/guardian satisfaction with pain control. If the parents/guardians cannot be reached by telephone, the participant's medical record will be reviewed to determine if there were any complications requiring a readmission to hospital. This phone call will take approximately 5-10 minutes to conduct each time. Following completion of the telephone call on day 14 following surgery, the child's participation in this study will be concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing coblation intracapsular tonsillectomy or adenotonsillectomy for sleep apnoea.
2. Between 3-9 years old (inclusive).
3. Patient(s) and guardian(s) can consent to participate in the study.
4. Legal guardian(s) can read and write in English.

Exclusion Criteria:

1. Patient or legal guardian refusal to participate in the study.
2. Emergency surgery.
3. Allergies to local anesthetics.
4. Patients with coagulopathy.
5. Congenital facial abnormalities including (but not limited to) hemifacial microsomia, maxillary hypoplasia, Treacher-Collins syndrome, and Goldenhar syndrome.
6. Developmental delay or neurological impairment including (but not limited to) Trisomy 21, cerebral palsy, and autism spectrum disorder.
7. Previous airway surgery or a known or predicted airway difficulty.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Impact of the suprazygomatic maxillary (SZMN) nerve block on opioid consumption in IV morphine equivalents in post-anesthesia care unit (PACU). | 0-24 hours following surgery
  This will be measured by evaluating the morphine consumption of participants during their time in the PACU and comparing the opioid requirements between study groups.

SECONDARY OUTCOMES:
Impact of the suprazygomatic maxillary (SZMN) nerve block on intraoperative and postoperative opioid consumption in IV morphine equivalents | During surgery - 14 days following surgery.
  This will be measured by evaluating participants' morphine consumption intraoperatively and postoperatively for 14 days following surgery and comparing the opioid requirements between study groups.
Impact of the suprazygomatic maxillary (SZMN) nerve block on postoperative pain scores | At completion of surgery - 14 days postoperative
  This will be measured by assessing patient pain scores using the FLACC (Face, Legs, Activity, Cry, Consolability) Pain Scale in the PACU and on days 1, 7 and 14 following surgery and comparing the results between study groups. The scale ranges from 0-10 with 0 indicating no pain (better outcome) and 10 indicating maximum pain (worse outcome).
Impact of the suprazygomatic maxillary (SZMN) nerve block on postoperative complications | At completion of surgery - 14 days postoperative
  This will be measured by recording the occurrence of postoperative complications such as nausea and vomiting, respiratory complications, surgical complications, and nerve block complications and comparing the results between study groups.
Impact of the suprazygomatic maxillary (SZMN) nerve block on the requirement for postoperative non-opioid analgesic consumption | At completion of surgery - 14 days postoperative
  This will be measured by evaluating the participants' consumption of non-opioid analgesics postoperatively for 14 days following surgery and comparing the results between study groups.
Impact of the suprazygomatic maxillary (SZMN) nerve block on the results of the Parental Satisfaction Questionnaire | At completion of surgery - 14 days postoperative
  This will be measured by the completion of the Parental Satisfaction Questionnaire that will be completed by the participants' parents/caregivers in the postoperative period to determine their satisfaction with their child's pain management and comparing the results between study groups. The Parental Satisfaction Questionnaire asks parents/guardians to assess certain aspects of their child's care to be either "positive" or "negative."
Impact of the suprazygomatic maxillary (SZMN) nerve block on the duration of participants'' stay in the post-anesthesia care unit (PACU) | Up to one day following surgery.
  This will be measured by recording the length of time participants are in the PACU and comparing the results between study groups.
Impact of the suprazygomatic maxillary (SZMN) nerve block on the results of the Postoperative Swallowing Assessment Scale | At completion of surgery - 14 days postoperative
  This will be measured by assessing the swallowing ability of participants using the Postoperative Swallowing Assessment Scale up to 14 days following surgery and comparing the results between study groups. The scale used to assess swallowing ability will range from 1-4 with 1 representing not being able to swallow (worse outcome) and 4 representing tolerating a regular diet with normal swallowing abilities (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Biswas, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lauder G, Emmott A. Confronting the challenges of effective pain management in children following tonsillectomy. Int J Pediatr Otorhinolaryngol. 2014 Nov;78(11):1813-27. doi: 10.1016/j.ijporl.2014.08.011. Epub 2014 Aug 27. PMID 25241379
- [Background] Alm F, Lundeberg S, Ericsson E. Postoperative pain, pain management, and recovery at home after pediatric tonsil surgery. Eur Arch Otorhinolaryngol. 2021 Feb;278(2):451-461. doi: 10.1007/s00405-020-06367-z. Epub 2020 Sep 26. PMID 32980893
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update). Otolaryngol Head Neck Surg. 2019 Feb;160(1_suppl):S1-S42. doi: 10.1177/0194599818801757. PMID 30798778
- [Background] Subramanyam R, Varughese A, Kurth CD, Eckman MH. Cost-effectiveness of intravenous acetaminophen for pediatric tonsillectomy. Paediatr Anaesth. 2014 May;24(5):467-75. doi: 10.1111/pan.12359. Epub 2014 Mar 5. PMID 24597962
- [Background] Brown KA, Laferriere A, Moss IR. Recurrent hypoxemia in young children with obstructive sleep apnea is associated with reduced opioid requirement for analgesia. Anesthesiology. 2004 Apr;100(4):806-10; discussion 5A. doi: 10.1097/00000542-200404000-00009. PMID 15087614
- [Background] Jensen DR. Pharmacologic management of post-tonsillectomy pain in children. World J Otorhinolaryngol Head Neck Surg. 2021 May 29;7(3):186-193. doi: 10.1016/j.wjorl.2021.03.004. eCollection 2021 Jul. PMID 34430826
- [Background] Lin C, Abboud S, Zoghbi V, Kasimova K, Thein J, Meister KD, Sidell DR, Balakrishnan K, Tsui BCH. Suprazygomatic Maxillary Nerve Blocks and Opioid Requirements in Pediatric Adenotonsillectomy: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Jul 1;150(7):564-571. doi: 10.1001/jamaoto.2024.1011. PMID 38780948
- [Background] Echaniz G, De Miguel M, Merritt G, Sierra P, Bora P, Borah N, Ciarallo C, de Nadal M, Ing RJ, Bosenberg A. Bilateral suprazygomatic maxillary nerve blocks vs. infraorbital and palatine nerve blocks in cleft lip and palate repair: A double-blind, randomised study. Eur J Anaesthesiol. 2019 Jan;36(1):40-47. doi: 10.1097/EJA.0000000000000900. PMID 30308523
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329